CLINICAL TRIAL: NCT01408524
Title: A Comparative Study in the Control of Emergence Blood Pressure During Craniotomy for Tumor Surgery Between Labetolol (Avexa) and Diltiazem
Brief Title: Control of Emergence Blood Pressure During Craniotomy for Tumor Surgery Between Labetolol and Diltiazem
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, busara sirivanasandha, Miss, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 594/2552(EC4)
Record Dates: First submitted 2011-07-11; First posted 2011-08-03 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension; Craniotomy
Keywords: Hypertension; emergence; craniotomy; Hypertension during the emergence after craniotomy
MeSH Terms: conditions — Hypertension | interventions — Diltiazem; Labetalol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diltiazem (Active Comparator): 2.5 mg iv q 2-5 min for keeping SBP below 140 mmHg during the emergence
  Interventions: Drug: Diltiazem
- Labetalol (Active Comparator): 2.5 mg iv q 2-5 min for keeping SBP below 140 mmHg during the emergence
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Diltiazem — 2.5 mg iv q 2-5 min for keeping SBP below 140 mmHg during the emergence
  Other Names: Herbessor
  Arms: Diltiazem
Drug: Labetalol — 2.5 mg iv q 2-5 min for keeping SBP below 140 mmHg during the emergence
  Other Names: Avexa
  Arms: Labetalol

SUMMARY:
The purpose of this study is to determine the effectiveness of the antihypertensive drugs in the control of emergence blood pressure after tumor resection craniotomy; compared between labetalol (Avexa) and diltiazem (Herbessor).

Also the investigators seek to determine the effective dose of the antihypertensive drugs and their side effects in Thai population.

DETAILED DESCRIPTION:
The study was randomized equivalence trial

ELIGIBILITY:
Inclusion Criteria:

* patients who scheduled for craniotomy for tomor removal

Exclusion Criteria:

* allergic to labetalol or diltiazem
* Bradycardia < 60 beat/min
* Second or third degree heart block
* Severe asthma or severe COPD
* Brain stem tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The number of the patients who have systolic blood pressure below 140 mmHg | 3 hours

SECONDARY OUTCOMES:
mean doses of the study drugs | 3hr
the number of patients with Adverse Events as a Measure of Safety and Tolerability | 6 hour

CONTACTS AND LOCATIONS:
Overall Officials: Busara - Sirivanasandha, MD, Principal Investigator — Department of Anesthesiology, Siriraj Hospital, Mahidol University, Bangkok, Thailand